CLINICAL TRIAL: NCT05117957
Title: Efficacy and Safety of Sorafenib in Previously Treated Advanced Hepatocellular Carcinoma: SOPT Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bo Hyun Kim (Other Government)
Responsible Party: Sponsor-Investigator, Bo Hyun Kim, Adjunct Associate Professor, Senior Scientist, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOPT study 2021
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: HCC; Sorafenib
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sorafenib (Experimental): Sorafenib will be administered orally at a dose of 600mg (3 tablets; 400mg orally in the morning and 200mg orally in the evening about 12 hours apart or 200mg orally in the morning and 400mg orally in the evening about 12 hours apart) daily without food (at least 1 hour before or 2 hours after a meal).
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Subjects will receive sorafenib 600mg orally daily. When dose reduction is necessary during the treatment of HCC, the sorafenib dose should be reduced to 400mg once daily. Escalation of sorafenib from a daily dose of 600mg to 800mg (400mg twice daily) is allowed if the subject who is tolerating the 600mg sorafenib dose level well. Treatment will continue until progression, unacceptable toxicity, withdrawal of consent, or study end, whichever occurs first.

SUMMARY:
To investigate the efficacy and safety of sorafenib administered as later lines of treatment in patients with advanced HCC.

DETAILED DESCRIPTION:
Sorafenib (Soranib Tablet) will be administered orally at a dose of 600mg daily without food for patients who have been treated with prior systemic therapy for advanced HCC. The study drug is continued until disease progression, unacceptable toxicity, withdrawal of consent, or study closure.

Response to sorafenib should be assessed at least every 8 weeks (± 7 days) by either CT scan or MRI.

After the treatment phase, subjects will undergo follow up for survival and the use of other anticancer treatments and/or therapies every 12 weeks (± 7 days) from the last dose and the survival follow up will be performed for at least 12 months after the enrollment of the last subject.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age of 20 or more
3. Histological or clinical diagnosis of HCC based on the guidelines of the Korean Liver Cancer Association-National Cancer Center
4. Locally advanced unresectable or metastatic disease not amenable to curative surgical and/or locoregional therapies
5. Intolerant to or progressed on at least 1 prior systemic treatment for HCC
6. Having at least one measurable target lesion (per RECIST v1.1)

   - Patients who received prior local therapy (e.g., radiofrequency ablation, transarterial chemoembolization, transarterial embolization, radiation therapy etc.) are eligible provided that other target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST 1.1.
7. Child-Pugh class A or B7
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
9. Life expectancy of at least 16 weeks
10. Adequate hematologic and hepatic function (should be obtained within 14 days prior to initiation of study treatment):
11. Women of childbearing potential and men must agree to use highly efficient contraception since signing of the IC form until at least 5 months (women) and 7 months (men) after the last study drug administration.

Exclusion Criteria:

1. Fibrolamellar carcinoma or sarcomatoid carcinoma
2. Having active brain metastasis or leptomeningeal metastasis
3. Moderate to severe or intractable ascites
4. Presence of hepatic encephalopathy
5. Presence of active bacterial infection
6. Uncontrolled severe medical comorbidity
7. Other malignant disease (a history of treated malignancy -other than HCC- is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding two years)
8. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Until 12 months after the last patient was enrolled
  Progression-free survival (PFS) is defined as the time from the date of treatment initiation to the date of the first observation of progressive disease (PD) by independent radiologic review according to RECIST criteria (version 1.1) or death from any cause.
Safety (Adverse events) | Until 12 months after the last patient was enrolled
  Incidence of adverse events will be evaluated.

SECONDARY OUTCOMES:
Overall survival (OS) | Until 12 months after the last patient was enrolled
  OS is defined as the time from the date of treatment initiation to the date of death.
Time to progression (TTP) | Until 12 months after the last patient was enrolled
  TTP is defined as the time from the date of treatment initiation to the date of the first observation of PD by independent radiologic review according to RECIST criteria (version 1.1).
Objective response rate (ORR) | Until 12 months after the last patient was enrolled
  ORR is defined as the proportion of enrolled subjects whose best overall response is a complete response (CR), or partial response (PR) using the RECIST criteria (version 1.1).
Disease control rate (DCR) | Until 12 months after the last patient was enrolled
  DCR is defined as the proportion of enrolled subjects whose best overall response is a CR or PR or stable disease (SD) using the RECIST criteria (version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Hyun Kim, M.D., Principal Investigator — National Cancer Center, South Korea
Locations (1):
- National Cancer Center, Korea, Seoul, South Korea